CLINICAL TRIAL: NCT06579820
Title: Effect of Tubular Bandage Application on Peripheral Intravenous Catheter Usage Time and Infiltration in Children
Acronym: chıldren
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, DİLEK SÖNMEZ SAĞLIK, principal investigator, Istanbul University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: DSONMEZSAGLIK
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Child, Only
Keywords: child, infiltration,catheter usage time

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group consisted of the group to which a tubular bandage was placed over the routinely applied peripheral intravenous catheters.
  Interventions: Combination Product: tubular bandage
- control group (No Intervention): The routine practice used for the application of peripheral intravenous catheters in the ward constituted the control group.

INTERVENTIONS:
Combination Product: tubular bandage — The experimental group consisted of the group in which a tubular bandage was applied over the PIC, which was routinely applied.
  Arms: experimental group

SUMMARY:
In pediatric patients, placement of peripheral intravenous catheters is the most commonly performed invasive medical procedure. In addition to the administration of medications, parenteral nutrition, intravenous fluids, and blood products, peripheral intravenous catheters are placed prophylactically before procedures and for emergency use in unstable patients.

One of the most common complications of peripheral intravenous catheters is infiltration. Infiltration is a vascular trauma resulting from a lesion in the vascular layers and subsequent perforation, resulting in the leakage of medications or non-vesicant solutions into the tissues surrounding the site of placement of the peripheral venous catheter.

In pediatric patients, physical factors (e.g. hyperactivity, sweating), tight fixation (may affect blood circulation and iatrogenic skin injury), loose fixation (may cause peripheral intravenous catheter displacement and infection), poor-quality fixation (may cause unplanned removal and skin injuries due to pressure), etc. causes more peripheral intravenous catheter fixation problems in pediatric patients than in adult patients Additional fixation products may be effective in preventing dislocation and micromotion in an active pediatric patient. However, limited recommendations regarding medical adhesive tapes and additional fixation products are guided only by low-evidence studies. The purpose of this study was to determine the effect of tubular bandage use on the duration of pediatric peripheral intravenous catheter use and the incidence of infiltration.

DETAILED DESCRIPTION:
RESEARCH OBJECTIVES AND DESIGN The study was conducted as a randomized controlled experimental design to determine the effect of tubular bandage application on the duration of peripheral venous catheter use and the frequency of infiltration in children aged 6-12 years who were receiving intravenous (I.V.) fluids through a peripheral venous catheter in the pediatric infection ward. RESEARCH HYPOTHESES Hypothesis 0 (H0): There is no significant effect of tubular bandage application on the duration of peripheral venous catheter use and the frequency of infiltration in children.

Hypothesis 1 (H1): The duration of peripheral venous catheter use is longer in children who receive tubular bandage application compared to those who do not. Hypothesis 2 (H2): The frequency of infiltration is lower in children who receive tubular bandage application compared to those who do not. RESEARCH VARIABLES The dependent variables of the study are the duration of peripheral venous catheter use and the frequency of infiltration occurrence. The independent variable is defined as tubular bandage application. RESEARCH POPULATION AND SAMPLE For this experimental study, the sample size was calculated as 100 participants in total (50 for each group) based on a power analysis derived from a similar study conducted by Atıcı et al. in 2019 with 49 patients. The randomization was done using the urn method, which is equivalent to full randomization. In the urn method, two parameters (α and β) are discussed, represented by two different colored balls: red and white. α can be either white or red, and β represents the ball of the opposite color to α. One ball is randomly selected, and if the selected ball is white, the individual is assigned to the α group, while if it is red, they are assigned to the β group. This process is repeated for each assignment. In the study, the red color was assigned to the experimental group, and the white color was assigned to the control group. When a child met the sampling criteria, these pre-prepared balls were placed in a black bag, and any nurse on duty was asked to select a ball with closed eyes. Based on the color of the selected ball, the child was assigned to either the control or experimental group, ensuring random distribution of participants into two groups. Sample Selection Criteria

* Willingness to participate in the study
* Parent/child's proficiency in Turkish
* Intact skin integrity in the application area
* First-time application of the peripheral venous catheter to the middle part of the child's forearm
* Recommendation by a physician for intravenous fluid containing 5% dextrose, 0.45% NaCl (sodium chloride), and 75% KCL(potassium chloride) through a peripheral venous catheter
* Child's age between 6-12 years
* Successful placement of the peripheral venous catheter on the first attempt

Sample Exclusion Criteria

* Coagulation abnormalities
* Receiving blood and blood products through the peripheral venous catheter
* Nutritional issues
* Hematologic or oncologic diseases
* Congenital genetic or neurological disorders
* Problems with skin integrity and movement in the upper extremities
* Sensitivity to the tubular bandage
* Fever above 37.5°C
* Accidental dislodgement of the catheter
* Early completion of treatment and removal of the catheter DATA COLLECTION FORMS AND TOOLS

The data collection process utilized the following:

* Data Collection Form
* Pediatric Peripheral Infusion Scale

The auxiliary tools used in data collection include:

* Tubular Bandage
* Transparent Adhesive Cove

ELIGIBILITY:
inclusion criteria

Willingness to participate in the study

* Parent/child's proficiency in Turkish
* Intact skin integrity in the application area
* First-time application of the peripheral venous catheter to the middle part of the child's forearm
* Recommendation by a physician for intravenous fluid containing 5% dextrose, 0.45% NaCl, and 75% KCL through a peripheral venous catheter
* Child's age between 6-12 years
* Successful placement of the peripheral venous catheter on the first attempt

exclusion criteria

Coagulation abnormalities

* Receiving blood and blood products through the peripheral venous catheter
* Nutritional issues
* Hematologic or oncologic diseases
* Congenital genetic or neurological disorders
* Problems with skin integrity and movement in the upper extremities
* Sensitivity to the tubular bandage
* Fever above 37.5°C
* Accidental dislodgement of the catheter
* Early completion of treatment and removal of the catheter

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
pediatric peripheral infiltration scale, information collection form | about a year
  The effect of tubular bandage on infiltration and catheter use time in children will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: dilek sönmez sağlık, Principal Investigator — dilek.sonmez@istanbul.edu.tr
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University, Istanbul, Fatih
  - Istanbul Unıversity, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsh N, Larsen EN, Takashima M, Kleidon T, Keogh S, Ullman AJ, Mihala G, Chopra V, Rickard CM. Peripheral intravenous catheter failure: A secondary analysis of risks from 11,830 catheters. Int J Nurs Stud. 2021 Dec;124:104095. doi: 10.1016/j.ijnurstu.2021.104095. Epub 2021 Sep 26. PMID 34689013
- [Background] Santos LMD, Conceicao TB, Silva CSGE, Tavares SS, Rocha PK, Avelar AFM. Care related to peripheral intravenous catheterism in pediatrics performed by nursing technicians. Rev Bras Enferm. 2021 Oct 18;75(2):e20200611. doi: 10.1590/0034-7167-2020-0611. eCollection 2021. English, Portuguese. PMID 34669898
- [Background] Ullman AJ, Takashima M, Kleidon T, Ray-Barruel G, Alexandrou E, Rickard CM. Global Pediatric Peripheral Intravenous Catheter Practice and Performance: A Secondary Analysis of 4206 Catheters. J Pediatr Nurs. 2020 Jan-Feb;50:e18-e25. doi: 10.1016/j.pedn.2019.09.023. Epub 2019 Oct 21. PMID 31648879
- [Background] Huang LS, Huang Y, Hu J. Current practices of peripheral intravenous catheter fixation in pediatric patients and factors influencing pediatric nurses' knowledge, attitude and practice concerning peripheral intravenous catheter fixation: a cross-sectional study. BMC Nurs. 2021 Nov 23;20(1):236. doi: 10.1186/s12912-021-00758-1. PMID 34814906
- [Background] Corley A, Ullman AJ, Mihala G, Ray-Barruel G, Alexandrou E, Rickard CM. Peripheral intravenous catheter dressing and securement practice is associated with site complications and suboptimal dressing integrity: A secondary analysis of 40,637 catheters. Int J Nurs Stud. 2019 Dec;100:103409. doi: 10.1016/j.ijnurstu.2019.103409. Epub 2019 Aug 28. PMID 31629208
- [Background] Corley A, Marsh N, Ullman AJ, Rickard CM. Peripheral intravenous catheter securement: An integrative review of contemporary literature around medical adhesive tapes and supplementary securement products. J Clin Nurs. 2023 May;32(9-10):1841-1857. doi: 10.1111/jocn.16237. Epub 2022 Feb 3. PMID 35118759
- [Background] Bahl A, Gibson SM, Jankowski D, Chen NW. Short peripheral intravenous catheter securement with cyanoacrylate glue compared to conventional dressing: A randomized controlled trial. J Vasc Access. 2023 Jan;24(1):52-63. doi: 10.1177/11297298211024037. Epub 2021 Jun 11. PMID 34112019
- [Background] Alexandrou E, Ray-Barruel G, Carr PJ, Frost SA, Inwood S, Higgins N, Lin F, Alberto L, Mermel L, Rickard CM; OMG Study Group. Use of Short Peripheral Intravenous Catheters: Characteristics, Management, and Outcomes Worldwide. J Hosp Med. 2018 May 30;13(5). doi: 10.12788/jhm.3039. PMID 29813140
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/ — pubmed